CLINICAL TRIAL: NCT07391566
Title: Phase 1b/2 Clinical Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of LPM6690176 Capsules in Combination With Chemotherapy and Bevacizumab in Metastatic Colorectal Cancer Patients With RAS Mutation
Brief Title: LPM6690176 in Combination With Chemotherapy and Bevacizumab in Metastatic Colorectal Cancer Patients With RAS Mutation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LY01024/CT-CHN-102
Record Dates: First submitted 2025-12-09; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LPM6690176 24 mg/m2 (Experimental): LPM6690176 capsules administered 24 mg/m2 orally Day 1 through Day 5 and Day 15 through Day 19 of each 28-day cycle in combination with FOLFIRI+Bevacizumab
  Interventions: Drug: LPM6690176; Biological: Bevacizumab; Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)
- LPM6690176 36 mg/m2 (Experimental): LPM6690176 capsules administered 36 mg/m2 orally Day 1 through Day 5 and Day 15 through Day 19 of each 28-day cycle in combination with FOLFIRI+Bevacizumab
  Interventions: Drug: LPM6690176; Biological: Bevacizumab; Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)
- LPM6690176 42 mg/m2 (Experimental): LPM6690176 capsules administered 42 mg/m2 orally Day 1 through Day 5 and Day 15 through Day 19 of each 28-day cycle in combination with FOLFIRI+Bevacizumab
  Interventions: Drug: LPM6690176; Biological: Bevacizumab; Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan)

INTERVENTIONS:
Drug: LPM6690176 — LPM6690176 orally.
Biological: Bevacizumab — Bevacizumab intravenously
Drug: FOLFIRI (5-Fluorouracil, Folinic acid, Irinotecan) — FOLFIRI intravenously

SUMMARY:
This study is consist of phase 1b (dose escalation + safety run-in) and phase 2 (randomized, controlled). Phase 1b is planned to evaluate the safety and tolerability of LPM6690176 capsule in combination with chemotherapy and Bevacizumab in patients with RAS mutant metastatic colorectal cancer (mCRC), to observe the dose-limiting toxicity (DLT), and to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D); Phase 2 is planned to preliminarily evaluate the efficacy of LPM6690176 capsule in combination with chemotherapy + Bev vs. chemotherapy + Bev in patients with previously untreated, RAS mutant mCRC.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed informed consent;
2. Age ≥ 18 years and ≤ 75 years, both male and female;
3. Histologically confirmed metastatic colorectal cancer (CRC) with RAS mutation;
4. Prior therapies for colorectal cancer:

(1 ) For phase 1b patients: who have failed or intolerable to prior first-line therapy; (2) For phase 2 patients: who have not received prior systemic therapy for metastatic colorectal cancer.

5. At least one measurable lesion according to RECIST 1.1 criteria; 6. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1; 7. Life expectancy≥ 6 months; 8. Adequate bone marrow and organ function; 9. Negative pregnancy test for women of childbearing potential. patients of childbearing potential should take effective contraceptive measures during study drug treatment and until 6 months after initiation of investigational product.

Exclusion Criteria:

1. Patients with known microsatellite instability (MSI-H) or mismatch repair deficiency (dMMR) who are suitable for immune checkpoint inhibitor therapy as assessed by the investigator;
2. Malignant tumors other than mCRC within 5 years before signing the informed consent;
3. Patients who did not recover from the AE of previous anti-tumor treatment to ≤ Grade 1;
4. Patients with body cavity effusion requiring local treatment or poorly controlled effusion;
5. Symptomatic brain metastasis, history of spinal cord compression or meningeal metastasis;
6. Underwent other therapeutic surgery other than diagnosis, biopsy, drainage, or expected to require major surgery during the study, or had unhealed wound, ulcer or fracture.
7. Current or previous uncontrolled concomitant non-gastrointestinal disease including, but not limited to myocardial infarction, unstable angina, coronary artery/peripheral artery bypass grafting, heart failure, cerebrovascular accident, transient ischemic attack, pulmonary embolism, deep vein thrombosis, serious arrhythmia, current uncontrolled hypertension, previous history of hypertensive crisis or hypertensive brain disease, tumor invasion into major blood vessels, interstitial lung disease, interstitial pneumonia, pulmonary interstitial fibrosis, reversible posterior leukoencephalopathy syndrome (RPLS), etc.;
8. Current or past presence of the gastrointestinal abnormalities, including but not limited to active peptic ulcer, clinically significant gastrointestinal abnormalities prior to informed consent, active colitis, long-term anticoagulant therapy, antiplatelet therapy, etc.;
9. Current or past significant risk of bleeding;
10. Use of prohibited medication or therapy within the specified time;
11. History of drug abuse or alcoholism;
12. Known hypersensitivity to any component of any investigational product;
13. Pregnant and lactating women;
14. Other conditions that may increase the risk of the study or interfere with study results, in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose-limiting toxicities (DLTs) | From the first dose of study drug treatment through Cycle 1 (28 days)
Phase Ib: Maximum tolerated dose (MTD) | From the first dose of study drug treatment through Cycle 1 (28 days)
Phase 1b: Recommended Phase 2 Dose (RP2D) | From the first dose of study drug treatment through Cycle 1 (28 days)
Phase 2: Overall response rate (ORR) | Approximately 2 years

SECONDARY OUTCOMES:
Phase 1b: Overall response rate (ORR) | Approximately 2 years
Duration of response (DOR) | Approximately 2 years
Disease control rate (DCR) | Approximately 2 years
Progression-free survival (PFS) | Approximately 2 years
Overall survival (OS) | Approximately 2 years
Maximum plasma concentration (Cmax) | From Pre-dose of Cycle 1 Day 1 and up to Cycle 1 Day 9 (Approximately 10 days, each cycle is 28 days)
Time to maximum plasma concentration (Tmax) | From Pre-dose of Cycle 1 Day 1 and up to Cycle 1 Day 9 (Approximately 10 days, each cycle is 28 days)
Area under the plasma concentration-time curve (AUC) | From Pre-dose of Cycle 1 Day 1 and up to Cycle 1 Day 9 (Approximately 10 days, each cycle is 28 days)
Elimination half-life (t1/2) | From Pre-dose of Cycle 1 Day 1 and up to Cycle 1 Day 9 (Approximately 10 days, each cycle is 28 days)
Trough observed plasma concentration (Ctrough) | From Pre-dose of Cycle 1 Day 1 and up to Cycle 1 Day 19 (Approximately 20 days, each cycle is 28 days)
Adverse Events (AEs) | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China